CLINICAL TRIAL: NCT01558193
Title: The Impact of Supplementation With Multi-vitamins/Minerals, With and Without Fatty Acids, on Impulsivity and Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Responsible Party: Principal Investigator, David Benton, Professor of Psychology, Swansea University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: DB-0123-DHAVM
Record Dates: First submitted 2012-02-28; First posted 2012-03-20 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Aggression
Keywords: Aggression DHA; Docosahexaenoic acid; Impulsivity; Minerals; Vitamins
MeSH Terms: conditions — Aggression; Impulsive Behavior | interventions — Geritol; Minerals; Docosahexaenoic Acids; efalex; Vitamins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Two placebos consumed
  Interventions: Dietary Supplement: Placebo
- Multi-vitamin/mineral (Active Comparator): Subjects took multi-vitamin/mineral and placebo fatty acid capsule
  Interventions: Dietary Supplement: Multi-vitamin/mineral
- Docosahexaenoic acid (Active Comparator): Subjects took docosahexaenoic acid capsule and placebo vitamins/minerals
  Interventions: Dietary Supplement: Docosahexaenoic acid
- DHA plus vitamins/minerals (Active Comparator): Subjects took both fatty acid and vitamin/mineral supplements
  Interventions: Dietary Supplement: DHA plus vitamins/minerals

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo for DHA of identical appearance - based on olive oil
  Placebo for vitamins/minerals of identical appearance
  Other Names: Does not apply
  Arms: Placebo
Dietary Supplement: Multi-vitamin/mineral — Each active tablet contained vitamins A (800µg); B1 (1.4mg); B2 (1.75mg); B6 (2mg); B12 (2.5mg); biotin 62.5 µg; folic acid 200 µg; niacin 20 mg; C (100mg); D (5µg); E (15mg); K (30µg); pantothenic acid (7.5 mg). In addition several minerals were administered: calcium (162mg); phosphorus (125mg); magnesium (100mg); potassium (40mg); chloride (36.3mg); iron (5mg); iodine (100µg); copper (500µg); manganese (2mg); chromium (40µg); molybdenum (50µg); selenium (30µg); zinc (5mg) as well as lutein (500 µg) . The placebo capsule was identical in color, size and appearance.
  Other Names: Centrum Advance 50+ (Pfizer Inc, New York)
  Arms: Multi-vitamin/mineral
Dietary Supplement: Docosahexaenoic acid — 22:6 (n-3) docosahexaenoic each capsule contained 224.2mg and three were taken per day
  Other Names: Efalex (Efamol Ltd, Leatherhead, England)
  Arms: Docosahexaenoic acid
Dietary Supplement: DHA plus vitamins/minerals — The DHA and vitamin/mineral supplements are as above
  Other Names: Efalex (Efamol Ltd); Centrum Advance 50+ (Pfizer Inc, New York)
  Arms: DHA plus vitamins/minerals

SUMMARY:
There is a series of well designed studies that have reported, in those with a history of anti-social behavior, that supplementation with vitamins / minerals, omega-3 fatty acids (n-3 FA), or both, reduces the incidence of aggressive behavior. Although there is evidence that all these nutrients have a role, to date the relative contribution of fatty acids and vitamins / minerals has not been considered: for example the possibility of a synergistic interaction has not yet been examined. In addition the topic has to date been studied under real-life condition, such as a prison, making the topic difficult to study. The major aim of the present study was to develop a paradigm that would allow the study of the topic in a sample from the general population without a history of anti-social behavior. Subjects received either a vitamin/mineral supplement, a fatty acid supplement, both or neither for three months, Measures of impulsivity and aggression were assessed before and after supplementation. Although in the past measures of actual behaviour have proved to be sensitive to supplementation, questionnaire measures have not. The second major objective was therefore to consider whether such phenomena can be studied in a sample without a history of anti-social behavior, using standardized, sensitive laboratory based measures and to compare these with questionnaire measures.

POLYMORPHISMS AND THE RESPONSE TO MICRO-NUTRIENT SUPPLLMENTATION The data set were subsequently used to test an a priori hypothesis not related to the initial hypothesis. A meta-analysis found a consistent pattern that micro-nutrient supplementation improved mood (Long SJ, Benton D. Effects of vitamin and mineral supplementation on stress, mild psychiatric symptoms, and mood in nonclinical samples: a meta-analysis. Psychosom Med 2013; 75: 144-153). To produce evidence of possible mechanisms the extent was determined, to which the impact of micro-nutrient supplementation was influenced by a range of polymorphisms associated with neurotransmitter systems known to modulate mood.

The primary outcome measure was the General Health Questionnaire, a 30-item self-report questionnaire that was developed to detect, in a community sample, those who would benefit from seeing a psychiatrist.

Given the literature that relates polymorphisms to mood disorders, and the known pharmacology of anti-depressant drugs, a range of polymorphisms were chosen associated with serotonin and catecholamines.

Dopamine The SNPs associated with the metabolism and functioning of dopamine were: Dopamine beta hydroxylase (DBH, rs16111115); Dopamine transporter (DAT1, rs2550946); Catechol-O-methyltransferase (COMT, rs4680, rs6269). Dopamine receptor D1 (DRD1, rs4532); Dopamine receptor D2 (DRD2, rs1079598, rs1800497); Dopamine receptor D3 (DRD3, rs6280); Dopamine receptor D4 (DRD4, rs1800955).

Serotonin Ten SNPs associated with different aspects of serotonin metabolism were also considered. Rs1843809 is a SNP of the TPH2 gene that encodes Tryptophan hydroxylase. Rs1050565 is a SNP in the BLMH gene that influences the activity of 5HTT (SLC6A4), the serotonin transporter. SNPs associated with various serotonin receptors were also examined: genetic variations of the HTR1A gene (5-HT1A receptor, rs6295); HTR1B gene (5-HT1B receptor, rs6296); HTR2A gene (5-HT2A receptor, rs6311); HTR2B gene (5-HT2B receptor, rs1549339); HTR2C gene (5-hydroxytryptamine receptor 2C, rs518147); HTR3A gene (5-hydroxytryptamine receptor 3A, rs1150226); HTR3B (5-HT3B receptor, rs1672717); HTR4 gene (5-HT4 receptor, rs2278392).

Adrenergic mechanisms Finally six SNPs associated with adrenergic receptors were considered: ADRA2A (adrenoceptor alpha 2A, rs553668); ADRB1 (adrenoceptor alpha B1, rs1801253); ADRB2 (adrenoceptor alpha B2, rs1042713; ADRB3 (adrenoceptor alpha B3, rs4994); SLC6AC (noradrenaline transporter, rs5569 and rs2242447).

Analysis The data will be analyzed using analysis of variance with a change in GHQ from before to after supplementation as the dependent variable: Micronutrient/placebo X Polymorphism.

DETAILED DESCRIPTION:
Objective: To consider whether aggression and impulsivity respond to multi-vitamins / minerals or fatty acid supplementation and whether there is a synergistic interaction?

In a between subjects design four groups will be contrasted. Those who for three months:

1. Receive two placebos
2. Receive multi-vitamin / mineral plus a placebo
3. Receive fatty acids plus placebo
4. Receive multi-vitamin / mineral plus fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Only male participants are being studied of self-reported good health who do not regularly consume seafood. They will be of a minimum age of 18 years of age and a maximum of 35 years of age. They will not be currently taking any medication and have no acute or chronic medical condition

Exclusion Criteria:

* If they had consumed n-3 fatty acid ro vitamin/mineral supplements during the previous six months.
* If they have any history of food intolerance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Go Stop Impulsivity Paradigm | Change from before to after supplementation for three months
  The GoStop Impulsivity Paradigm measures the ability to inhibit an already initiated response. A number of five digits are presented on a computer screen for 500ms followed by a 500ms blackout. A second number then appears for 500ms followed by a 500ms blackout. If the numbers are identical the mouse button has to be pressed before the second number disappeared. However, the response has to be with-held if a "Stop" signal appeared; that is the second number was identical but changed from black to red. If the two numbers were different then no response was required.
Rosenzweig Picture Frustration Test | Change from before to after supplementation for three months
  This is test of the tendency to respond in an aggressive manner. A series of cartoons are presented that present an intentionally frustrating situation. The participant reports what he or she would say in that situation. Blind the responses are assessed in terms of the extent to which the responses are aggressive in matter
  Note that the use of two primary outcomes reflects the aim of the study to contrast performance and questionnaire measures

SECONDARY OUTCOMES:
Buss Perry Aggression Scale | Change from before to after supplementation for three months
  The Buss-Perry Aggression Questionnaire assesses four aspects of aggressive behavior: physical aggression, verbal aggression, anger and hostility. Participants rank statements about their temperament using a 7-point Likert scale ranging from 1 (extremely uncharacteristic of me) to 7 (extremely characteristic of me).
Perceived Stress Scale | Change from before to after supplementation for three months
  The Perceived Stress Scale assesses the extent to which stressful thoughts and feeling had been experienced during the last month. For example: "In the last month, how often have you been upset because of something that happened unexpectedly?" The participant responded on a scale ranging from 0 = Never to 4 = Very Often. An overall score is calculated.
Single Key Impulsivity Paradigm | Change from before to after supplementation for three months
  A measure of the subjects ability to forgo initial reward for a later larger reward. The subject can choose to wait for a reward and get more points or alternatively respond more quickly and get fewer points sooner. The longer a subject waits the higher the reward; that the more points are earned. A mouse click began the task and a second resulted in a reward. Two counters display the most recent and cumulative reward over a 20 minute session. Subject are able to infer that responses at a faster rate earn smaller rewards.
General Health Questionnaire | Further analysis of existing data - considers changes from baseline to three months
  Polymorphisms associated with the metabolism and receptors of dopamine and serotonin will be related to the response to micro-nutrient supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David Benton, D.Sc, Principal Investigator — Swansea University, Swansea, United Kingdom, SA2 8PP
Locations (1):
- Swansea University, Swansea, Wales, United Kingdom